CLINICAL TRIAL: NCT03584256
Title: Vitamin D Status Relate to Bone Mineral Density, Body Composition and Variey Cardiovascular Risk Factors Among Competitive Female Gymnasts and Swimmers After Winter Time
Brief Title: Vitamin D Status Among Competitive Female Gymnast and Swimmers After Winter Time
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Collaborators: Barbara Jakše s.p. (Other)
Responsible Party: Sponsor
Other Study IDs: 0120-177/2018
Record Dates: First submitted 2018-05-23; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Vitamin D Deficiency; Injuries; Cardiovascular Risk Factor; Nutritional Deficiency
MeSH Terms: conditions — Vitamin D Deficiency; Wounds and Injuries; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gymnasts: Female gymnasts, older than 13 years, with status of ineternational or national level,
- swimmers: Female swimmers, older than 12 years, with status of ineternational or national level,

SUMMARY:
As indoor athletes, competitive gymnasts and swimmers can face the problem of a potential vitamin D deficiency. In the last decades, indoor sports participants have been faced with the problem of an institutionalized lifestyle and, in some places, a lower exposure to sun, which is also associated with the geographical area with a lower or higher UV index, especially in autumn, winter, and early spring (from October to April), when the day is shorter and the clock shifts to winter time. The problem with gymnasts and swimmers lies in daily trainings in the gym and pool and in the daily rest between two trainings, which can be spend more or less institutionally. The investigators wanted to examine the vitamin D status related to bone mineral density, body composition and various cardiovascular markers among young competitive gymnasts and swimmers after winter time. The investigators want to potentially give more solid but sensible recommendations for trainers, athletes, parents and sports doctors when it comes to vitamin D supplementations for indoor female athletes.

DETAILED DESCRIPTION:
In this cross-sectional survey, the investigators will document vitamin D and the status of other micronutrients related to bone mineral density, body composition and a variety of risk factors for chronic non-communicable diseases.

The investigators hypothesize that there exists a serious problem of vitamin D deficiency among indoor athletes related to bone health, injuries and general health - especially when they are not using supplements. It is well known that vitamin D may improve athletic performance in vitamin D-deficient athletes.

International and national-level female gymnasts and swimmers that will be enrolled will sign an informed consent statement for the inclusion in this survey and the choice to participate in the study will be made by coaches and participants themselves and, in the event of females under 18 years of age, also by their parents, in accordance with the Helsinki declaration.

The investigators plan to enroll at least 30 female participants (15 gymnasts and 15 swimmers) who compete on an international and national level and are older than 12 years of age.

The investigators will measure the athletes' biochemistry in overnight fasted state (micronutrients, including vitamin D (25(OH)D), B12, Ca, Fe, Mg, K and P, lipids, liver enzymes, glucose, creatinine, etc.), their seated blood pressure status, bone mineral density (also segmental) and body composition, using Dual-energy X-ray absorptiometry (DXA), their dietary choice and nutrition intake status, using standardized Food frequency questionnaire (FFQ), their training characteristics, injury status and menstrual status. Athletes who are using vitamin D supplements or who have attended a one-month training camp in the southern geographical zone (Africa) will serve us as control group.

ELIGIBILITY:
Inclusion Criteria:

* international and national level
* Signed informed consent for participation in the study

Exclusion Criteria:

-

Min Age: 12 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Sport
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Differences between female gymnasts and swimmers of vitamin D status | April 2018
  Serum 25(OH)D (ng/ml) status after winter time

SECONDARY OUTCOMES:
Differences between female gymnasts and swimmers of bone mineral density status | April 2018
  Bone mineral density status (g/cm3) using DEXA

OTHER OUTCOMES:
Differences between female gymnasts and swimmers of body composition status | April 2018
  Lean and fat tissue mass (%) assessed dy DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Čuk, Principal Investigator — University of Ljubljana, Faculty of Sport, Slovenia
Locations (1):
- Faculty of Sport, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bjelakovic G, Gluud LL, Nikolova D, Whitfield K, Wetterslev J, Simonetti RG, Bjelakovic M, Gluud C. Vitamin D supplementation for prevention of mortality in adults. Cochrane Database Syst Rev. 2014 Jan 10;2014(1):CD007470. doi: 10.1002/14651858.CD007470.pub3. PMID 24414552
- [Background] Fuleihan Gel-H, Bouillon R, Clarke B, Chakhtoura M, Cooper C, McClung M, Singh RJ. Serum 25-Hydroxyvitamin D Levels: Variability, Knowledge Gaps, and the Concept of a Desirable Range. J Bone Miner Res. 2015 Jul;30(7):1119-33. doi: 10.1002/jbmr.2536. Epub 2015 May 7. PMID 25952470
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Bannert N, Starke I, Mohnike K, Frohner G. [Parameters of mineral metabolism in children and adolescents in athletic training]. Kinderarztl Prax. 1991 May;59(5):153-6. German. PMID 1921165
- [Background] Lovell G. Vitamin D status of females in an elite gymnastics program. Clin J Sport Med. 2008 Mar;18(2):159-61. doi: 10.1097/JSM.0b013e3181650eee. PMID 18332692
- [Background] De Keyzer W, Dekkers A, Van Vlaslaer V, Ottevaere C, Van Oyen H, De Henauw S, Huybrechts I. Relative validity of a short qualitative food frequency questionnaire for use in food consumption surveys. Eur J Public Health. 2013 Oct;23(5):737-42. doi: 10.1093/eurpub/cks096. Epub 2012 Jul 26. PMID 22843611
- [Background] Geiker NRW, Hansen M, Jakobsen J, Kristensen M, Larsen R, Jorgensen NR, Hansen BS, Bugel S. Vitamin D Status and Muscle Function Among Adolescent and Young Swimmers. Int J Sport Nutr Exerc Metab. 2017 Oct;27(5):399-407. doi: 10.1123/ijsnem.2016-0248. Epub 2017 May 30. PMID 28556690
- [Derived] Jakse B, Jakse B, Cuk I, Sajber D. Body Composition, Training Volume/Pattern and Injury Status of Slovenian Adolescent Female High-Performance Gymnasts. Int J Environ Res Public Health. 2021 Feb 19;18(4):2019. doi: 10.3390/ijerph18042019. PMID 33669675